CLINICAL TRIAL: NCT04774484
Title: Impact of High-Intensity Interval Training on Regulatory T Cells
Brief Title: High-Intensity Interval Training and Regulatory T Cells
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not available.
Sponsor: Francesc Marti (Other)
Responsible Party: Sponsor-Investigator, Francesc Marti, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2020-10-11; First posted 2021-03-01 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: End Stage Renal Disease
Keywords: high intensity; interval training; exercise; obesity; inflammation; Treg
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity; Obesity; Inflammation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects will be in one arm (Experimental): Both Lean and Obese, End-Stage Renal Disease (ESRD) patients and normal volunteers will be in one arm, that will receive the High Intensity Interval Training intervention.
  Interventions: Other: High Intensity Interval Training

INTERVENTIONS:
Other: High Intensity Interval Training — After the acclimatization session and assessment of eligibility, a graded exercise test (GXT) will be given to the participant. After checking their vitals, the HIIT program will be performed on recumbent cycles. The first two weeks of training will consist of a gradual ramp where subjects will perform a moderate intensity cycling program consisting of a 5-minute warm up followed by progressively longer continuous cycling starting at 15 minutes and progressing up to 30 minutes prior to starting the HIIT training. For the HIIT training subjects will perform 5 minutes of low to moderate steady state cycling to warm up. Following the warm up, the subjects will complete the 4x4 HIIT program. This will consist of 4 minutes of cycling at 85% of the subject's maximum heart rate (HR) followed by 4 minutes of a low intensity cycling period for recovery.

SUMMARY:
Regulatory T cells (Tregs) are a small population of T cells compromising of 1% to 5% of the total T cells in the body but they are playing a fundamental role in the maintenance of the immune homeostasis. These cells modulate the immune system by suppressing the effector activity and thus preventing autoimmune diseases and chronic inflammatory processes. Treg cell numbers have shown to increase with physical activity, and this increment has been directly correlated with exercise intensity. These results suggest that the increased Treg frequency may contribute to the beneficial effects of exercise on disorders associated with autoimmune disease or chronic low-grade inflammation such as atherosclerosis, diabetes mellitus, chronic kidney disease or cancer.

The overall purpose of this study is to determine the influence High-intensity interval training (HIIT) on the frequency and quality of peripheral Treg cells.

DETAILED DESCRIPTION:
Tregs have been studied in clinical practice for different therapeutic applications. In the past several years there has been a significant interest in the transplant community to develop tolerance in order to substantially decrease or even eliminate the need of immuno-suppressive regimens. A growing body of evidence recognizes the balance between graft-reactive effector cells and graft-protective suppressor Treg cells as the ultimate determinant of long-term allograft survival. As a result, there is a major interest in transplantation to enhance the suppressor immune response as an alternative or complementary approach to reach a clinical tolerogenic state and preserve graft function. Exercise improves baseline immune function and helps to maintain immune homeostasis. Treg cell numbers have shown to increase with physical activity, and this increment has been directly correlated with exercise intensity. These results suggest that the increased Treg frequency may contribute to the beneficial effects of exercise on disorders associated with autoimmune disease or chronic low-grade inflammation such as atherosclerosis, diabetes mellitus, chronic kidney disease or cancer.

Primary Objectives: The overall purpose of this study is to determine the influence High-intensity interval training (HIIT) on the frequency and quality of peripheral Treg cells.

Secondary Objectives: Effects of HIIT in other T cell populations. Effects of HIIT in plasma concentration of inflammatory and metabolic markers. Effects of HIIT in obese vs lean.

Design: This is a prospective, single center, single-arm "pre-test/post-test" study designed to evaluate the safety, feasibility and initial efficacy of a 12-week HIIT regimen to increase the frequency and quality of peripheral Treg cells. All participants will have a pre-test (baseline) evaluation followed by a treatment and then a post-test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old.
* BMI between 18.5 and 25 or above 30. Rationale: we want to include "obesity" as categorical covariate in the influence of HIIT and discriminate the participants between "lean" (BMI range 18.5-25) and "obese" (BMI > 30)
* Sedentary lifestyle (fewer than 5,000 steps per day)
* Fluent in English, able to understand and provide informed consent.
* Subjects willing to participate in the study and comply with study requirements as evidenced by signed Institutional Review Board (IRB)-approved informed consent.

Exclusion Criteria:

* Age under 18 or over 65
* BMI under 18.5 or between 25 and 30.
* Active lifestyle (more than 5,000 steps per day).
* Previous chronic use of systemic glucocorticoids, immune-suppressors or immuno-modulators in the preceding 3 months.
* Patients with significant or active infection: HIV negative by ELISA or reverse transcription polymerase chain reaction (RT-PCR) [if ELISA is positive and RT-PCR is negative, the ELISA is considered false positive]; negative serology for Hepatitis B and C.
* Active malignancy or history of malignancy within 1 year.
* Be pregnant or breastfeeding.
* Hemoglobin less than 9.0 g/dl at the time of blood drawing.
* Platelet count less than 100,000/* at the time of blood drawing.
* White blood count less than 4 and/or Absolute Neutrophil Count less than 1500/* at the time of blood drawing.
* Participation in any other study that involved investigational drug or regimens in the preceding 12 months.
* History of delayed or abnormal wound healing.
* Any immuno-related condition, chronic illness or prior treatment which, in the opinion of the investigator, precludes study participation.
* Inability or unwillingness of participant to comply with study protocol or procedures.
* Impaired consent capacity.
* Any chronic use of anticoagulation.
* Recipient of blood transfusion in 3 months prior to blood drawing.
* Any orthopedic condition or chronic pain that prevents them from cycling.
* Any symptomatic coronary artery disease prior enrollment within 3 months or any intervention for it in the past 6 months.
* Any symptomatic current heart failure (New York Heart Association class III and IV), significant valvar heart disease.
* History of non-compliance.
* The study will not include any vulnerable population such as fetuses, pregnant women, children, or prisoners.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline concentration of circulating Regulatory T cells (Tregs) in blood at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of circulating Regulatory T cells (Tregs) in blood
Change from baseline Serum C-Reactive protein at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Adiponectin at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline expansion rates of TRegs (in vitro) at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline expansion rates of TRegs

SECONDARY OUTCOMES:
Change from baseline Serum Interleukin-6 (IL6) at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Tumor Necrosis Factor- Alpha (TNF-alpha) at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Leptin at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Blood Glucose at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Triglycerides at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Total Cholesterol at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Low Density Lipoprotein (LDL) at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline High Density Lipoprotein (HDL) at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Insulin at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Intracellular Helios at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Cell membrane CD36 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Cell membrane GLUT1 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Cell membrane Leptin-Receptor at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Cell membrane TIGIT at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Suppressor Activity at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline activty of the Functional activity of TRegs
Change from baseline Intracellular FoxP3 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Membrane CD25 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker
Change from baseline Membrane CD127 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the Treg phenotype marker

OTHER OUTCOMES:
Change from baseline Serum IL10 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Interferon Gamma (IFNg) at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Epinephrine at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum NorEpinephrine at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Serum Lactate at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline concentration of serologic cytokines/growth factors/metabolites
Change from baseline Intracellular Eomes at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Intracellular RORyt at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Intracellular Tbet at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane OX40 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane GITR at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker ofTreg cells
Change from baseline Cell membrane DR3 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane 41BB at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CCR2 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CCR4 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CCR6 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CCR7 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CXCR3 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CD226 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Intracellular CTLA4 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane ICOS at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane PD1 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane PDL1 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CD39 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane CD49d at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Cell membrane LAP-T at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Intracellular Granzyme-Beta at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker ofTreg cells
Change from baseline Intracellular IL35 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline Intracellular IL10 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of Treg cells
Change from baseline TSRD-Met at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Changes from baseline methylation status of tsrd promoter - Treg lineage commitment
Change from baseline Intracellular Tbet at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of conventional-Effector TH1 T cells
Change from baseline Intracellular IFNg at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of conventional-Effector TH1 T cells
Change from baseline Intracellular GATA3 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of conventional-Effector TH2 T cells
Change from baseline Intracellular IL5 at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of conventional-Effector TH2 T cells
Change from baseline Intracellular RORgt at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of conventional-Effector TH17 T cells
Change from baseline Intracellular IL17af at 12 weeks post HIIT intervention | Baseline- and at 12 weeks post-HIIT intervention
  Change from baseline percentage and intensity of the phenotype marker of conventional-Effector TH17 T cells

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Marti, PhD, Principal Investigator — University of Kentucky, College of Medicine / Transplant Center
Locations (1):
- University of Kentucky Transplant Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No